CLINICAL TRIAL: NCT07017361
Title: A Multicenter Randomized Prospective Study on Establishing an ERAS Program and Optimized Clinical Protocol for Patients Undergoing Minimally Invasive Pancreatoduodenectomy (MIPD)
Brief Title: ERAS Program Implementation for MIPD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: SMG-SNU Boramae Medical Center (Other); Korea University Anam Hospital (Other)
Responsible Party: Principal Investigator, Wooil Kwon, Associate Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-2502-154-1619
Record Dates: First submitted 2025-05-20; First posted 2025-06-12 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Pancreaticoduodenectomy; ERAS; Minimally Invasive Surgery
Keywords: Pancreaticoduodenectomy; ERAS; Minimally Invasive Surgery
MeSH Terms: interventions — Congresses as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional (Active Comparator)
  Interventions: Procedure: Conventional
- ERAS (Experimental)
  Interventions: Procedure: ERAS

INTERVENTIONS:
Procedure: Conventional — Pre-operative fasting: NPO for solids and fluids from 00:00. No pre-emptive oral analgesia. Intra-operative: IV dexamethasone 5 mg at anaesthesia induction; IV acetaminophen 1 g about 1 h before wound closure. Post-operative nutrition: Levin tube removed in OR. POD1 morning-sips of water; POD3 morning upright abdominal X-ray; if normal, start soft fluid diet POD3 evening. POD4 pancreatobiliary CT; if normal, start soft bland diet at lunch. Drain management: two drains at hepaticojejunostomy and pancreaticojejunostomy; drain amylase measured POD1, 3 and 5; if POD4 CT normal, drains removable from POD5 per surgeon discretion (output, fever, pain). Analgesia: IV PCA until ≈POD3, then oral acetaminophen 650 mg every 8 h. No carbohydrate loading or NSAID/nefopam adjuncts.
  Arms: Conventional
Procedure: ERAS — Pre-op fasting: solids NPO from 00:00; clear fluids until 3 h pre-op; 300 mL carbohydrate drink 2-4 h pre-op with oral acetaminophen 650 mg + zaltoprofen 80 mg. Intra-op: IV dexamethasone 8 mg at induction; IV acetaminophen 1 g + ibuprofen 300 mg + nefopam 20 mg 1 h before closure. Post-op nutrition: Levin tube removed in OR. POD1 sips of water; POD2 morning upright abdominal X-ray-if normal, start soft fluid diet POD2 evening. POD3 pancreatobiliary CT-if normal, start soft bland diet at lunch. Drain mgmt: same placement; amylase POD1 & 3; if POD4 CT normal and amylase ≤ 5 000 U/L trending down, remove drains POD4; otherwise per surgeon. Analgesia: IV PCA until ≈POD3; until POD1 morning, IV acetaminophen 1 g + ibuprofen 300 mg q8h; POD1-5, oral acetaminophen 650 mg + zaltoprofen 80 mg q8h.
  Arms: ERAS

SUMMARY:
To evaluate the impact of an Enhanced Recovery After Surgery (ERAS) program on postoperative recovery in patients undergoing minimally invasive pancreatoduodenectomy (MIPD)

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 19 years, scheduled for standard minimally invasive (robotic or laparoscopic) pancreatoduodenectomy for periampullary tumors
* ECOG performance status of 0 or 1 at screening
* Able to provide written informed consent, understand study procedures, and complete patient-reported questionnaires
* ASA physical status classification I-III

Exclusion Criteria:

* Hypersensitivity to fentanyl or ropivacaine
* Cognitive impairment preventing independent use of patient-controlled analgesia or completion of questionnaires
* Major internal medical or psychiatric disorders affecting treatment response
* Severe hepatic or renal dysfunction
* Any condition deemed inappropriate for study participation by the investigator

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-07-15 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants Meeting Discharge Criteria by Post-operative Day 5 Afternoon | Up to the afternoon of Post-operative Day 5

SECONDARY OUTCOMES:
Length of Post-operative Hospital Stay (Days) | Post-operative Day 0 until hospital discharge (assessed up to Post-operative Day 30)
Incidence of Major Complications (Clavien-Dindo ≥ Grade IIIa) Within 30 Days | Post-operative Day 0 to Day 30
Total Direct Medical Costs per Participant (KRW) During Index Hospitalization | Post-operative Day 0 until hospital discharge (assessed up to Post-operative Day 30)

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Daehak-ro, Jongno-gu, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-06-03): https://cdn.clinicaltrials.gov/large-docs/61/NCT07017361/Prot_SAP_000.pdf